CLINICAL TRIAL: NCT05063045
Title: Development and Preliminary Effects of Smart Cloth Care System for Persons With Dementia
Brief Title: Smart-Cloth Care System for Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MOST 107-2314-B-182-007
Record Dates: First submitted 2021-09-15; First posted 2021-09-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Dementia, Senile; Family Members
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A quasi-experimental design using experimental and control group but without random assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart-cloth (Experimental): Participants receive smart-cloth assisted home nursing care
  Interventions: Behavioral: smart-cloth assisted home nursing care
- routine care (No Intervention): This group receive routine care

INTERVENTIONS:
Behavioral: smart-cloth assisted home nursing care — Older persons with dementia or hip fracture were asked to wear a smart vest, which contained a coin-size monitor in a hidden inner pocket. Sensors were installed in bedrooms and living areas to receive signals from the smart clothing. The home care nurses then gave feedback from the sensor signals to family caregivers.
  Arms: smart-cloth

SUMMARY:
The purpose of this study is to develop and examine the preliminary effects of a smart cloth care system for facilitating family caregiving for persons with dementia in the home setting. This will be a three-year study, with the first two years to explore the feasibility of such a smart cloth care system and the third year to pilot test its effects. During the third year, a quasi experimental design will be implemented and the outcomes of caregivers and persons with dementia will be followed for 6 months.

DETAILED DESCRIPTION:
The purpose of this study is to develop and examine the preliminary effects of a smart cloth care system for facilitating family caregiving for persons with dementia in the home setting. A smart-care model, using smart clothing with a remote monitoring system, was developed to assist home-nursing care. Older persons with dementia are asked to wear a smart vest, which contained a coin-size monitor in a hidden inner pocket. Sensors are installed in bedrooms and living areas to receive signals from the smart clothing. Alarm at door, emergency button and smoke detector are also installed. The signals and emergency information are transmitted to the mobile phones of responsible home care nurses, who have downloaded an app to their phones. After the home care nurse receive a sensor signal, she would then give feedback to family caregivers about the care receiver, including emergency calls, frequent getting up at night, staying in the bathroom for more than 30 minutes, inadequate or abnormal activity level, not moving during the day for more than 2 hours, leaving the house alone, and a sensor being disconnected from the system. Based on information and signals from smart-care sensors, home care nurses will discuss caregiving activities and planning with family caregivers.Participants were asked to wear smart clothing for at least 4 days/week for 6 months. A home care research nurse will visit the home setting to assess it for sensor installation and suggest environmental modifications for potential hazards. A second visit will be made by an engineer with the research nurse to install the sensors. The research nurse visit the participants' homes once a week during the first month and once every month from the second to third month after the sensor installation to conduct in-home interventions and resolve problems using the smart-care system.

During the first two years, this smart cloth care system will be developed. During the third year. The investigators plan to recruit at least 60 participants and randomize them into an intervention group (N=30) that receives the smart cloth care model and a control group (N=30) that receives usual care. Patient and caregiver outcomes will be followed every two months for a period of 6 months after the smart cloth care system has been implemented. Finally Intention-to-treat and hierarchical linear models will be used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

Older persons were included by these criteria:

age 60 or older diagnosed with dementia, or received surgery for a hip fracture could walk independently or with assistance living with family members in northern Taiwan.

Family caregivers were included by these criteria:

* 20 years old responsible for providing direct care or supervising care received by the patient.

Exclusion Criteria:

Terminal ill Living in institution

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Time UP and Go | two months after installation
  Time spends while stand from an armed chair, walk for three meters and come back to sit down
Time UP and Go | four months after installation
  Time spends while stand from an armed chair, walk for three meters and come back to sit down
Time UP and Go | six months after installation
  Time spends while stand from an armed chair, walk for three meters and come back to sit down
Barthel Activity of Daily Living Scale | two months after installation
  dependency in activities of daily living, 0-100, higher score indicate better activities of daily living.
Barthel Activity of Daily Living Scale | four months after installation
  dependency in activities of daily living, 0-100, higher score indicate better activities of daily living.
Barthel Activity of Daily Living Scale | six months after installation
  dependency in activities of daily living, 0-100, higher score indicate better activities of daily living.
IADL self-care ability | two months after installation
  dependency in instrumental activities of daily living
IADL self-care ability | four months after installation
  dependency in instrumental activities of daily living
IADL self-care ability | six months after installation
  dependency in instrumental activities of daily living
cognitive function | two months after installation
  Mini-Mental State Examination
cognitive function | four months after installation
  Mini-Mental State Examination
cognitive function | six months after installation
  Mini-Mental State Examination
Medical Outcome Short Form-36 | two months after installation
  Health-related quality of life, from 0-100, higher score representing better health related quality of life
Medical Outcome Short Form-36 | four months after installation
  Health-related quality of life, from 0-100, higher score representing better health related quality of life
Medical Outcome Short Form-36 | six months after installation
  Health-related quality of life, from 0-100, higher score representing better health related quality of life
Preparedness scale | two months after installation
  caregiver preparedness for caregiving, 10-50, higher score indicate better preparedness
Preparedness scale | four months after installation
  caregiver preparedness for caregiving, 10-50, higher score indicate better preparedness
Preparedness scale | six months after installation
  caregiver preparedness for caregiving, 10-50, higher score indicate better preparedness
Centre for epidemiological Studies Depression Scale | two months after installation
  caregiver depressive symptoms, 0-60, higher score indicate more depressive symptoms
Centre for epidemiological Studies Depression Scale | four months after installation
  caregiver depressive symptoms, 0-60, higher score indicate more depressive symptoms
Centre for epidemiological Studies Depression Scale | six months after installation
  caregiver depressive symptoms, 0-60, higher score indicate more depressive symptoms
caregiver balance scale | two months after installation
  caregiving balance between competing needs, 0-3, higher score indicate more balanced
caregiver balance scale | four months after installation
  caregiving balance between competing needs, 0-3, higher score indicate more balanced
caregiver balance scale | six months after installation
  caregiving balance between competing needs, 0-3, higher score indicate more balanced
Caregiver Medical Outcome Short Form-36 | two months after installation
  caregiver health-related quality of life, from 0-100, higher score representing better health related quality of life
Caregiver Medical Outcome Short Form-36 | four months after installation
  caregiver health-related quality of life, from 0-100, higher score representing better health related quality of life
Caregiver Medical Outcome Short Form-36 | six months after installation
  caregiver health-related quality of life, from 0-100, higher score representing better health related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ing L Shyu, PhD, Principal Investigator — School of Nursing, Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Taiwan, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sung YL, Huang HL, Lin CC, Kroger T, Hsu WC, Hsu JL, Lin YE, Shyu YL. Experiences of family caregivers of persons living with dementia with and without a smart- clothes assisted home nursing program during the heightened COVID-19 alert. BMC Geriatr. 2022 Aug 23;22(1):697. doi: 10.1186/s12877-022-03379-8. PMID 35996089